CLINICAL TRIAL: NCT06018376
Title: Characteristics of Sexual Dysfunction in Patients With Lung Cancer
Acronym: LUDICAS
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 23/01_LUDICAS
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Sexual Dysfunction
Keywords: Lung Cancer; Sexual Dysfunction
MeSH Terms: conditions — Lung Neoplasms; Sexual Dysfunction, Physiological | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study Group: * Age greater than or equal to 18 years and less than or equal to 70 years.
  * Diagnosis of lung cancer stages IB to IV.
  * Having received systemic oncological treatment for at least 3 months
  * ECOG ≤ 2
  Interventions: Drug: Systemic oncological treatment

INTERVENTIONS:
Drug: Systemic oncological treatment — Oncological systemic treatment for at least 3 months or being in oncological follow-up after having received systemic treatment for a minimum of 3 months
  Other Names: chemotherapy; radiotherapy

SUMMARY:
The general objective of this observational study is identify and describe the type, frequency, and severity of sexual dysfunction in patients with lung cancer and generate strategies for clinical management and oncological follow-up directed and based on the specific findings in this population. The recruitment will be carried out from July 2023 and will be carried out until December 2023, the analysis of the information will be carried out from January to March 2024.

DETAILED DESCRIPTION:
It is planned to develop a study with a larger number of patients with lung cancer, including the population of Spain and Latin American countries to obtain a sample of more diverse and heterogeneous characteristics, with clinical, cultural, and sociodemographic differences. This will make it possible to obtain better and greater data and therefore define the clinical and treatment factors significantly associated with DS in these individuals and obtain a more complete vision of the reality of the problem.

The results of this research will make it possible to carry out interventions specifically directed at this population and to modify the oncological follow-up guidelines currently in force. Likewise, the information collected will serve as the basis for generating new protocols for a multidisciplinary approach, including the participation of psychology and specialists in urology, gynecology, and psychiatry.

The general objective of this observational study is identify and describe the type, frequency, and severity of sexual dysfunction in patients with lung cancer and generate strategies for clinical management and oncological follow-up directed and based on the specific findings in this population. The recruitment will be carried out from July 2023 and will be carried out until December 2023, the analysis of the information will be carried out from January to March 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years and less than or equal to 70 years.
* Diagnosis of lung cancer stages IB to IV.
* Having received systemic oncological treatment for at least 3 months or being in oncological follow-up after having received systemic treatment for a minimum of 3 months with stable tumor disease or partial or complete response in images.
* ECOG ≤ 2

Exclusion Criteria:

* Patients with comorbidities (renal failure, cardiovascular diseases or similar) not controlled with corresponding medical management.
* Individuals with physical disability or cognitive impairment that prevents them from completing the electronic data collection form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer stages IB to IV with ECOG ≤ 2 between 18 and 70 years old that received systemic oncological treatment for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aylen Vanessa Ospina Serrano, MD, Study Chair — Hospital Puerta del Hierro Investigator
Locations (29):
- Instituto Alexander Flemming, Buenos Aires, Buenos Aires, Argentina
- Colombia (5):
  - Clínica Universitaria Colombia, Bogotá, Bogota D.C.
  - Clinica del Occidente, Cali, Cali
  - Hematooncologos SA, Cali, Cali
  - Clínica de Medellín, Medellín, MEdellín
  - Oncomedica, IMAT, Montería, Monteria
- ALIADAS Instituto Nacional de Enfermedades Neoplasicas, Surquillo, Perú, Peru
- Centro Hospitalar do Porto, Porto, Porto District, Portugal
- Spain (21):
  - Hospital General de Elche, Elche, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Hospital Universitari Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Xarxa sanitaria Santa Tecla- Tarragona, Tarragona, Tarragona
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Universitario Cruces, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ospina-Serrano AV, Maximiano C, Cantos B, Torrente M, Mendez M, Sanchez JC, Calvo V, Collazo-Lorduy A, Blanco M, Nunez B, Triana I, Parejo C, Martinez P, Duma N, Provencio-Pulla M. Sexual dysfunction in patients with cancer, a challenge in oncology practice: results of the CLARIFY project. Clin Transl Oncol. 2024 May;26(5):1147-1156. doi: 10.1007/s12094-023-03332-0. Epub 2023 Nov 2. PMID 37917247
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational Study Group
Started | 553
Completed | 448
Not Completed | 105

BASELINE CHARACTERISTICS:
Arm/Group | Observational Study Group
Number analyzed (Participants) | 448
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 277
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Spain | 408
  Colombia | 18
  Argentina | 14
  Portugal | 8
Smoking status [Count of Participants; unit: Participants]
  Smoker | 256
  Former smoker | 114
  Never smoker | 75
  Unknown | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.44 (7.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Different Type, Frequency and Severity of Sexual Dysfunction
Description: Identify and describe the type, frequency, and severity of sexual disfunction in patients with lung cancer and generate strategies for clinical management and oncological follow-up directed and based on the specific findings in this population.
Time Frame: From inclusion up to 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Female Participants: Females that met the follwing criteria:
  * Age greater than or equal to 18 years and less than or equal to 70 years.
  * Diagnosis of lung cancer stages IB to IV.
  * Having received systemic oncological treatment for at least 3 months
  * ECOG ≤ 2
- Male Participants: Males that met the following criteria:
  * Age greater than or equal to 18 years and less than or equal to 70 years.
  * Diagnosis of lung cancer stages IB to IV.
  * Having received systemic oncological treatment for at least 3 months
  * ECOG ≤ 2
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 171 | 277
Participants
  Severe Disturbances in sexual response phases: Desire | 71 | 275
  Severe Disturbances in sexual response phases: Arousal | 76 | 51
  Severe Disturbances in sexual response phases_ Orgasm | 70 | 71

ADVERSE EVENTS:
Time Frame: In this study, adverse events were not collected; therefore, there are no results available
Description: In this study, adverse events were not collected; therefore, there are no results available. Patients affected and patients at risk have been considered as "0" since no data is available.
Groups:
- Observational Study Group: In this study, adverse events were not reported; therefore, there are no results available
Arm/Group | Observational Study Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT06018376/Prot_SAP_000.pdf